CLINICAL TRIAL: NCT00201864
Title: Phase II Trial of Exemestane (Aromasin) in Combination With Fulvestrant (Faslodex) in Postmenopausal Women With Hormone Sensitive Advanced Breast Cancer
Brief Title: Exemestane in Combination With Fulvestrant in Postmenopausal Women With Hormone Sensitive Advanced Breast Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Ohio State University Comprehensive Cancer Center (Other)
Collaborators: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: OSU-0494; NCI-2011-03154 (Registry Identifier: Clinical Trial Reporting Program (CTRP))
Record Dates: First submitted 2005-09-12; First posted 2005-09-20 (Estimated); Results first posted 2016-08-15 (Estimated); Last update posted 2018-07-26 (Actual); Status verified 2018-06

CONDITIONS: Breast Cancer
Keywords: Postmenopausal; Women
MeSH Terms: conditions — Breast Neoplasms | interventions — exemestane; Fulvestrant

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- single-arm study (Experimental): Combination of daily exemestane 25 mg with monthly 250 mg Fulvestrant injection
  Interventions: Drug: Exemestane; Drug: Fulvestrant

INTERVENTIONS:
Drug: Exemestane — 25 mg orally per day
  Other Names: Aromasin
Drug: Fulvestrant — 250 mg IM starting on Day 8 and then every 28 days.
  Other Names: Faslodex

SUMMARY:
The purpose of this trial is to evaluate time to progression in women with hormone responsive advanced breast cancer treated with a combination of exemestane and fulvestrant.

ELIGIBILITY:
Inclusion Criteria:

* Proven breast cancer
* Metastatic or locally advanced breast cancer
* Hormonally responsive disease defined as estrogen (ER) and/ or progesterone receptor (PR) positive (>10% staining by immunohistochemistry)
* Postmenopausal status
* No more than 1 prior chemotherapy for stage IV metastatic breast cancer allowed
* ECOG (Eastern Cooperative Oncology Group) performance status 0-2
* Adequate organ function
* Exclusion Criteria:
* No prior Exemestane or Fulvestrant
* Uncontrolled intercurrent illness including but not limited to:

  * ongoing or active infection
  * symptomatic congestive heart failure
  * unstable angina pectoris
  * cardiac arrhythmia
  * myocardial infarction within the last 3 months
  * psychiatric illness/social situations that would limit compliance with study
* Lymphangitic pulmonary disease; carcinomatous meningitis, bone marrow only metastases; and a rising tumor marker without any other site of metastatic disease.
* Presence of bleeding diathesis or coagulopathy, patients requiring coumadin

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2005-09; Primary Completion 2012-06 (Actual); Study Completion 2014-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ewa Mrozek, MD, Principal Investigator — Ohio State University
Locations (1):
- Ohio State University, Columbus, Ohio, United States

REFERENCES:
- [Result] Mrozek E, Layman R, Ramaswamy B, Schaaf L, Li X, Ottman S, Shapiro CL. Phase II trial of exemestane in combination with fulvestrant in postmenopausal women with advanced, hormone-responsive breast cancer. Clin Breast Cancer. 2012 Apr;12(2):151-6. doi: 10.1016/j.clbc.2012.01.003. PMID 22444722
- See also: Jamesline — http://cancer.osu.edu

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients were enrolled between November 2005 and December 2009
Groups:
- Exemestane and Fulvestrant: Combination of daily exemestane 25 mg with monthly 250 mg Fulvestrant injection
  Exemestane: 25 mg orally per day
  Fulvestrant: 250 mg IM starting on Day 8 and then every 28 days.
Period: Overall Study
Arm/Group | Exemestane and Fulvestrant
Started | 40
Completed | 40
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Exemestane and Fulvestrant
Number analyzed (Participants) | 40
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 29
  >=65 years | 11
Age, Continuous [Median (Full Range); unit: years] | 58 [43 to 84]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 40
  Male | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 40
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 4
  White | 36
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 40
Time From Primary Diagnosis to Metastatic Disease [Median (Full Range); unit: years] | 5 [0 to 21]
Relapse and/or Progression [Number; unit: participants]
  During adjuvant endocrine therapy | 14
  >12 mo after completion adjuvant therapy | 9
  Presenting with de novo metastatic disease | 8
  Never on adjuvant hormonal therapy | 9

OUTCOME MEASURES:

1. Primary Outcome: Time to Progression (TTP) in Women With Hormone Responsive Advanced Breast Cancer Treated With Combination of Exemestane and Fulvestrant.
Description: TTP is defined as the time from first treatment to objective evidence of progression on the basis of radiological evaluation and/or physical exam (if physical examination identifies a site of measurable disease). Progression is defined using Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.0), as a 20% increase in the sum of the longest diameter of target lesions, or a measurable increase in a non-target lesion, or the appearance of new lesions
Time Frame: Every 2 cycles up to 2 years
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Exemestane and Fulvestrant
Number analyzed (Participants) | 40
months | 6.9 [3.9 to 13.5]

2. Secondary Outcome: Overall Clinical Benefit (Complete Response Rate, Partial Response and Stable Disease)
Description: Response and progression was evaluated after every 2 cycles by physical examination and imaging studies using the international RECIST criteria.
  Complete Response (CR), Partial Response (PR), Overall Response Rate (ORR), Stable Disease (SD), Progressive Disease (PD). Per Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.0) for target lesions and assessed by MRI and/or CT: Partial Response (PR), >=30% decrease in the sum of the longest diameter of target lesions; Stable Disease (SD), neither sufficient shrinkage to qualify for a Partial Response nor sufficient increase to qualify for Progressive Disease (PD); PD, 20% increase in the sum of the longest diameter of target lesions, or a measurable increase in a non-target lesion, or the appearance of new lesions; Complete Response (CR), Disappearance of all target lesions; Overall Response Rate (ORR), CR+PR
Time Frame: Every 2 cycles, up to 1 year
Measure: Number; unit: patients
Arm/Group | Exemestane and Fulvestrant
Number analyzed (Participants) | 40
patients
  CR | 0
  PR | 3
  ORR | 3
  SD ≥ 6 Mo | 17
  Overall Clinical Benefit | 20
  SD< 6 Mo | 8
  PD | 12

3. Secondary Outcome: Maximum Plasma Concentration (Cmax) of Exemestane When Administered Alone and With Fulvestrant
Description: 5 mL of venous whole blood was obtained before dosing and then at 1, 2, 4, 6, 8, and 24 hours after exemestane ingestion on each of the 2 time points.
Time Frame: Day 7 and Day 120
Population: Only 9 patients had evaluable PK data collected and analyzed
Measure: Mean (Standard Deviation); unit: ng/ml
Arm/Group | Exemestane and Fulvestrant
Number analyzed (Participants) | 9
ng/ml
  Exemestane Alone (Day 7) | 20.1 (7.7)
  Exemestane + Fulvestrant (Day 120) | 21.2 (11.1)
Statistical Analysis 1: Comparison: Exemestane and Fulvestrant; Test type: Superiority or Other; p = 0.9102, Wilcoxon (Mann-Whitney)

4. Secondary Outcome: Examine the Effect of Exemestane + Fulvestrant on Serum IGF-1 and IGFPB-3 Levels
Time Frame: Prestudy, Day 7 and Day 120
Population: Increase in mean levels from baseline to day 120. Not all patients had the IGF-1 and IGFBP-3 levels present.
Measure: Mean (Standard Deviation); unit: ng/mL
Groups:
- IGF-1: IGF-1-insulin-like growth factor
- IGFBP-3: IGFBP-3-insulin-like growth factor-binding
Arm/Group | IGF-1 | IGFBP-3
Number analyzed (Participants) | 23 | 22
ng/mL
  Baseline | 119 (41.1) | 4946 (1188)
  Day 7 | 141 (55.1) | 5273 (1372)
  Day 120 | 161 (61.2) | 5537 (1166)

ADVERSE EVENTS:
Description: The NCI Common Terminology Criteria for Adverse Events (CTCAE) v3.0 was used to assess adverse events for patients on this trial. The CTCAE using is a descriptive terminology that utilizes Adverse Event (AE) reporting.
Arm/Group | Single-arm Study
Serious Adverse Events (participants affected / at risk) | 6/40
Other Adverse Events (participants affected / at risk) | 24/40
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Single-arm Study (N=40)
Chest pain (General disorders) | 1 (1)
Thromboembolism (Vascular disorders) | 2 (2)
Nausea (Gastrointestinal disorders) | 1 (1)
Vomiting (Gastrointestinal disorders) | 1 (1)
Hypercalcemia (Metabolism and nutrition disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 3% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Single-arm Study (N=40)
Neutropenia (Blood and lymphatic system disorders) | 1 (1) — Grade 2 according to NCI Common Terminology Criteria for Adverse Events (CTCAE v.3.0)
Anemia (Blood and lymphatic system disorders) | 4 (4) — Grade 2 and Grade 3 according to NCI Common Terminology Criteria for Adverse Events (CTCAE version 3.0)
Thrombocytopenia (Injury, poisoning and procedural complications) | 2 (2) — Grade 2 according to NCI Common Terminology Criteria for Adverse Events (CTCAE version 3.0)
Fatigue (General disorders) | 14 (14) — Grade 2 and Grade 3 according to NCI Common Terminology Criteria for Adverse Events (CTCAE version 3.0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 6 (6)
Nausea (Gastrointestinal disorders) | 4 (4)
Vomiting (Gastrointestinal disorders) | 4 (4)
Anorexia (Metabolism and nutrition disorders) | 6 (6)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Bone pain (Musculoskeletal and connective tissue disorders) | 10 (10)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes